CLINICAL TRIAL: NCT04424199
Title: The Relationship Between Our Ability in Travelling in Time and in Estimating Time Duration and Their Interaction With Spatial Attention: a Neuropsychological Study.
Brief Title: Temporal Disorders in Left and Right Brain-Damaged Patients
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ICS Maugeri CE 2194-Ob1
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Brain Disease
Keywords: Time perception; Mental Time Travel; Prismatic adaptation; Left and Right Brain Damaged Patients
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- LBD patients R-PA: A group of 10 left brain damaged (LBD) patients will attend two sessions:
  1. First session - before prismatic adaptation (pre-PA): they will perform a computerized test battery to measure time abilities (Mental Time Travel and Time Estimation) and a neuropsychological test battery to assess cognitive abilities.
  2. Second session - after prismatic adaptation (post-PA): they will perform the Mental Time Travel and Time Estimation tasks immediately after a single session of pointing with prismatic goggles inducing rightward attentional shift (R-PA).
  Interventions: Behavioral: Rightward Attentional Shift (R-PA)
- LBD patients L-PA: A group of 10 left brain damaged (LBD) patients will attend two sessions:
  1. First session - before prismatic adaptation (pre-PA): they will perform a computerized test battery to measure time abilities (Mental Time Travel and Time Estimation) and a neuropsychological test battery to assess cognitive abilities.
  2. Second session - after prismatic adaptation (post-PA): they will perform the Mental Time Travel and Time Estimation tasks immediately after a single session of pointing with prismatic goggles inducing leftward attentional shift (L-PA).
  Interventions: Behavioral: Leftward Attentional Shift (L-PA)
- RBD patients R-PA: A group of 10 right brain damaged (RBD) patients will attend two sessions:
  1. First session - before prismatic adaptation (pre-PA): they will perform a computerized test battery to measure time abilities (Mental Time Travel and Time Estimation) and a neuropsychological test battery to assess cognitive abilities.
  2. Second session - after prismatic adaptation (post-PA): they will perform the Mental Time Travel and Time Estimation tasks immediately after a single session of pointing with prismatic goggles inducing rightward attentional shift (R-PA).
  Interventions: Behavioral: Rightward Attentional Shift (R-PA)
- RBD patients L-PA: A group of 10 right brain damaged (RBD) patients will attend two sessions:
  1. First session - before prismatic adaptation (pre-PA): they will perform a computerized test battery to measure time abilities (Mental Time Travel and Time Estimation) and a neuropsychological test battery to assess cognitive abilities.
  2. Second session - after prismatic adaptation (post-PA): they will perform the Mental Time Travel and Time Estimation tasks immediately after a single session of pointing with prismatic goggles inducing leftward attentional shift (L-PA).
  Interventions: Behavioral: Leftward Attentional Shift (L-PA)
- HC R-PA: A group of 10 healthy controls (HC) will attend two sessions:
  1. First session - before prismatic adaptation (pre-PA): they will perform a computerized test battery to measure time abilities (Mental Time Travel and Time Estimation) and a neuropsychological screening (Mini Mental State Examination) to assess inclusion/exclusion criteria.
  2. Second session - after prismatic adaptation (post-PA): they will perform the Mental Time Travel and Time Estimation tasks immediately after a single session of pointing with prismatic goggles inducing rightward attentional shift (R-PA).
  Interventions: Behavioral: Rightward Attentional Shift (R-PA)
- HC L-PA: A group of 10 healthy controls (HC) will attend two sessions:
  1. First session - before prismatic adaptation (pre-PA): they will perform a computerized test battery to measure time abilities (Mental Time Travel and Time Estimation) and a neuropsychological screening (Mini Mental State Examination) to assess inclusion/exclusion criteria.
  2. Second session - after prismatic adaptation (post-PA): they will perform the Mental Time Travel and Time Estimation tasks immediately after a single session of pointing with prismatic goggles inducing leftward attentional shift (L-PA).
  Interventions: Behavioral: Leftward Attentional Shift (L-PA)

INTERVENTIONS:
Behavioral: Rightward Attentional Shift (R-PA) — Patients will perform a session of 90 pointing movements toward a visual target presented on the right, the left or at the center of the visual field. This pointing task will be performed with prismatic googles inducing a rightward attentional shift.
  Groups: HC R-PA; LBD patients R-PA; RBD patients R-PA
Behavioral: Leftward Attentional Shift (L-PA) — Patients will perform a session of 90 pointing movements toward a visual target presented on the right, the left or at the center of the visual field. This pointing task will be performed with prismatic googles inducing a leftward attentional shift.
  Groups: HC L-PA; LBD patients L-PA; RBD patients L-PA

SUMMARY:
Time is an important function that permeates our everyday activities but it has been so far significantly under-investigated in neurological patients.

For instance, it is known that right brain damaged (RBD) patients with spatial attentional deficit (neglect) are impaired in both the ability to estimate the duration of an event (Time Estimation), showing a time underestimation, and the ability of mentally moving in past and future time (Mental Time Travelling), showing a deficit in processing future events when they are projected in the past. After a leftward shift of spatial attention induced by prismatic adaptation (PA), both the underestimation and the ability to travel in time ameliorate. However, less is known about these abilities in left brain damaged (LBD) patients.

Aims of this study are to investigate:

i) the performance (in terms of accuracy and reaction times) of LBD and RBD patients on Mental Time Travelling; ii) the correlation between Mental Time Travelling and Time Estimation abilities; iii) the efficacy of a single session of PA inducing a leftward (L-PA) and a rightward (R-PA) attentional shift on Mental Time Travelling and Time Estimation abilities.

A group of control subjects will be involved for comparison among groups.

DETAILED DESCRIPTION:
Time processing involves different abilities - i.e. estimating the duration of an event (Time Estimation) and moving in past and future time (Mental Time Travelling) - and it is a fundamental ability in everyday life. However, in neuropsychology, time processing is routinely neglected in the assessment of cognitive deficits in brain-damaged patients. This is surprising since time is an important function that permeates our activities: it is involved in perceiving mismatches in lip reading (milliseconds), estimating how long it takes to be ready for work (minutes), and planning how long it will take a manuscript to be accepted (usually months). Thus, impairment in processing time has important consequences in daily life.

For instance, it is known that right brain damaged (RBD) patients with spatial attentional deficit (neglect) underestimate durations of milliseconds and show a deficit in processing future events when they are projected in the past.

Moreover, previous studies have demonstrated that a leftward shift of spatial attention induced by prismatic adaptation (PA) determines an amelioration of both, time underestimation and the deficit in mental travel in time.

The Mental Time Travelling, in particular, seems to involve different cognitive functions, among others, episodic memory and the ability to anticipate the future. Recent evidence suggests that these functions are mediated by neural circuits localized in the left hemisphere but no studies have investigated the ability of mentally moving in past and future time in left brain damaged (LBD) patients.

Aims of this study are to investigate:

i) the performance (in terms of accuracy and reaction times) of LBD and RBD patients on Mental Time Travelling; ii) the correlation between Mental Time Travelling and Time Estimation abilities; iii) the efficacy of a single session of PA inducing a leftward (L-PA) and a rightward (R-PA) attentional shift on Mental Time Travelling and Time Estimation abilities.

A group of control subjects will be involved for comparison among groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with focal (right or left) brain-damage

Exclusion Criteria:

* generalized cognitive impairment (score lower than 24 at the Mini Mental State Examination)
* psychiatric disorders
* additional neurological disorders
* abusive use of alcohol or illicit drugs

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from primary care clinic and they will be compared with matched healthy controls. Healthy controls will be selected from a community sample who volunteer to participate in the research.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Change in Mental Time Travel Ability on the Mental Time Travel (MTT) Task | pre-PA and immediately post-PA
  In the MTT task participants are listened to auditory stimuli consisting of brief descriptions of personal and non-personal events. They are required to project themselves in the past (10 years ago), present or future (10 years from now) and to verbally determine whether each event has already happened (relative past event) or is yet to happen (relative future event) with respect to the specific self-location in time (past, present and future).
  Error rates and reaction times will be recorded and analyzed. The improvement will be defined as changes in the Inverse Efficiency (IE) ability: reaction times/accuracy.
Change in Time Estimation Ability on the Time Estimation Task | pre-PA and immediately post-PA
  The Time Estimation task consists of a red square that is displayed for different durations (1400, 1700, 2000, 2300, 2600 ms) on the computer screen. Participants are instructed to verbally judge whether the duration of each stimulus is "short" or "long" with respect to previously acquired pair of reference durations (1400 and 2600 ms).
  A psychophysical response function will be created for each participant by calculating the proportion of "long" responses: the Point of Subjective Equality (PSE) is the duration at which a participant is equally likely to classify the stimuli as short or long. An increase of "long" response after treatment, as compared to baseline performance, induces a decreased PSE, reflecting a relative shift towards overestimation of temporal midpoint. Conversely, an increase of "short" responses after treatment, as compared to baseline performance, induces an increased PSE, reflecting a relative shift towards underestimation of temporal midpoint.

SECONDARY OUTCOMES:
Assessment of Unilateral Spatial Neglect on the Behavioral Inattention Test (BIT) | baseline
  The BIT is composed of two scales, the Conventional scale and the Behavioral scale. Participants will be administered the Conventional scale, which includes 6 tasks: line crossing, letter cancellation, star cancellation, figure and shape copying, line bisection and representational drawing. The score ranges from 0 to 146 (cut-off = 129).
Assessment of Unilateral Spatial Neglect on the Bells Cancellation Test | baseline
  The subject is required to cross out the bells that are scattered among several different shapes on a sheet of paper. Two indices of neglect will be calculated: total number of omissions (cut-off < 5) and number of left omissions (cut-off < 5), i.e. the difference between the number of targets crossed out on the right side and the number of targets crossed out on the left side (asymmetry score).
Assessment of Unilateral Spatial Neglect on the Apples Cancellation Test | baseline
  This is a cancellation task in which outline drawings of 150 apples are shown pseudorandomly scattered over a sheet of A4 paper presented in a landscape orientation. All of the apples are presented in an upright position. One-third of the apples are full (targets) and two-thirds are open on either the left or the right side (distractors). Participants are asked to cross out all the full apples and to ignore the distractors. Three scores will be calculated: full apples barrage (cut-off = 45), full apples asymmetry (cut-off = 2), and incomplete apples asymmetry (cut-off = 1).
  The full apples asymmetry (the difference between the number of targets selected on the right side and the number of targets selected on the left side) represents the score for egocentric neglect. The incomplete apples asymmetry (total left openings minus total right openings) represents the score for allocentric neglect.
Assessment of General Cognitive Functioning on the Mini Mental State Examination (MMSE) | baseline
  The MMSE is a 30-point questionnaire that examines functions including registration (repeating named prompts), attention and calculation, recall, language, ability to follow simple commands and orientation. The score ranges from 0 to 30 (cut-off = 24).
Assessment of Verbal Comprehension on the Token Test | baseline
  The Token test is a test of auditory language processing in which participants are asked to manipulate tokens of different shapes, sizes, and colors in response to increasingly complex instructions. One point is credited for a correct performance on the first presentation and 0.5 point if the performance is correct only on the second presentation. The score ranges from 0 to 36 (cut-off = 26,50).
Assessment of Frontal Functions on the Frontal Assessment Battery (FAB) | baseline
  The FAB is a brief battery of six neuropsychological tasks designed to assess frontal lobe function at bedside. The six tasks explore: conceptualization and abstract reasoning, lexical verbal fluency and mental flexibility, motor programming and executive control of action, self-regulation and resistance to interference, inhibitory control, and environmental autonomy.
  Each task scores from 0 (pathologic) to 3 (best performance), for a total maximum score of 18.
Assessment of Memory on the Rey's 15 Words Auditory Learning Test | baseline
  The test is designed as a list-learning paradigm in which the participant hears a list of 15 nouns and is asked to recall as many words from the list as possible (five repetitions of free-recall). After a 15 min delay, the participant is asked to again recall the words from the list. It provides two scores: immediate (range 0-75) and delayed recall (range 0-15), i.e. the higher the score, the better the performance.
Assessment of Ideomotor Apraxia on the Movement Imitation Test | baseline
  The ability to carry out movements on imitation is assessed with a 24-item test. Each movement is presented for a maximum of 3 times and scores from 0 (pathologic) to 3 (best performance). The total score ranges from 0 to 72 (cut-off = 62).
Assessment of Verbal Estimation Ability on the Time and Weight Estimation Test (STEP) | baseline
  The STEP assesses aspects of executive functioning related to cognitive estimation ability. The questionnaire is composed of two distinct ten-item sections, focusing on time (e.g., How long does it take to have a shower?) and weight (e.g., How heavy is a pair of jeans?) estimations. Each item scores from 0 (bizarre estimation) to 3 (best estimation), for a total maximum score for each section of 30, with a cut-off value for normality above 20 for each section.
Assessment of Verbal Estimation Ability on the Cognitive Estimation Task (CET) | baseline
  The test comprised 21 questions that required participants to give oral, numerical responses. Two different scoring procedures will be considered: absolute error score and bizarreness. The total score for all 21 items ranges from a best of zero to a worst of 42. The greater the error score, the poorer the performance on the CET (cut-off = 18). The total bizarreness score ranges from 0 and 21 (cu-off = 4). The higher the bizarreness score, the greater the impairment in cognitive estimation.
Correlation between Time Processing Abilities | baseline
  MTT and Time Estimation Task will be correlated to investigate the relationship between different time processing abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Frassinetti, PhD, Principal Investigator — Istituti Clinici Scientifici Maugeri IRCCS
Locations (1):
- ICS Maugeri IRCCS, U.O. di Rieducazione e Recupero funzionale di Castel Goffredo, Castel Goffredo, Mantova, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anelli F, Avanzi S, Arzy S, Mancuso M, Frassinetti F. Effects of spatial attention on mental time travel in patients with neglect. Cortex. 2018 Apr;101:192-205. doi: 10.1016/j.cortex.2018.01.012. Epub 2018 Feb 2. PMID 29482017
- [Background] Anelli F, Avanzi S, Damora A, Mancuso M, Frassinetti F. Mental time travel and functional daily life activities in neglect patients: Recovery effects of rehabilitation by prism adaptation. Cortex. 2019 Apr;113:141-155. doi: 10.1016/j.cortex.2018.12.003. Epub 2018 Dec 14. PMID 30660953
- [Background] Appollonio I, Leone M, Isella V, Piamarta F, Consoli T, Villa ML, Forapani E, Russo A, Nichelli P. The Frontal Assessment Battery (FAB): normative values in an Italian population sample. Neurol Sci. 2005 Jun;26(2):108-16. doi: 10.1007/s10072-005-0443-4. PMID 15995827
- [Background] Bertossi E, Aleo F, Braghittoni D, Ciaramelli E. Stuck in the here and now: Construction of fictitious and future experiences following ventromedial prefrontal damage. Neuropsychologia. 2016 Jan 29;81:107-116. doi: 10.1016/j.neuropsychologia.2015.12.015. Epub 2015 Dec 18. PMID 26707714
- [Background] Bertossi E, Tesini C, Cappelli A, Ciaramelli E. Ventromedial prefrontal damage causes a pervasive impairment of episodic memory and future thinking. Neuropsychologia. 2016 Sep;90:12-24. doi: 10.1016/j.neuropsychologia.2016.01.034. Epub 2016 Jan 28. PMID 26827916
- [Background] Carlesimo GA, Caltagirone C, Gainotti G. The Mental Deterioration Battery: normative data, diagnostic reliability and qualitative analyses of cognitive impairment. The Group for the Standardization of the Mental Deterioration Battery. Eur Neurol. 1996;36(6):378-84. doi: 10.1159/000117297. PMID 8954307
- [Background] De Renzi E, Faglioni P. Normative data and screening power of a shortened version of the Token Test. Cortex. 1978 Mar;14(1):41-9. doi: 10.1016/s0010-9452(78)80006-9. PMID 16295108
- [Background] De Renzi E, Motti F, Nichelli P. Imitating gestures. A quantitative approach to ideomotor apraxia. Arch Neurol. 1980 Jan;37(1):6-10. doi: 10.1001/archneur.1980.00500500036003. PMID 7350907
- [Background] Della Sala S, MacPherson SE, Phillips LH, Sacco L, Spinnler H. How many camels are there in Italy? Cognitive estimates standardised on the Italian population. Neurol Sci. 2003 Apr;24(1):10-5. doi: 10.1007/s100720300015. PMID 12754651
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Mancuso M, Rosadoni S, Capitani D, Bickerton WL, Humphreys GW, De Tanti A, Zampolini M, Galardi G, Caputo M, De Pellegrin S, Angelini A, Bartalini B, Bartolo M, Carboncini MC, Gemignani P, Spaccavento S, Cantagallo A, Zoccolotti P, Antonucci G. Italian standardization of the Apples Cancellation Test. Neurol Sci. 2015 Jul;36(7):1233-40. doi: 10.1007/s10072-015-2088-2. Epub 2015 Jan 25. PMID 25618236
- [Background] Oliveri M, Magnani B, Filipelli A, Avanzi S, Frassinetti F. Prismatic adaptation effects on spatial representation of time in neglect patients. Cortex. 2013 Jan;49(1):120-30. doi: 10.1016/j.cortex.2011.11.010. Epub 2011 Nov 27. PMID 22200531
- [Background] Patane I, Farne A, Frassinetti F. Prismatic Adaptation Induces Plastic Changes onto Spatial and Temporal Domains in Near and Far Space. Neural Plast. 2016;2016:3495075. doi: 10.1155/2016/3495075. Epub 2016 Feb 14. PMID 26981286
- [Background] Wilson B, Cockburn J, Halligan P. Development of a behavioral test of visuospatial neglect. Arch Phys Med Rehabil. 1987 Feb;68(2):98-102. PMID 3813864